CLINICAL TRIAL: NCT02931487
Title: Restoring Emotion Regulation Networks in Depression Vulnerability: An Experimental Study Applying an Attention Bias Modification Procedure
Brief Title: Restoring Emotion Regulation Networks in Depression Vulnerability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Nils Inge Landrø, Professor Dr. philos, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HSØ-2015052
Record Dates: First submitted 2016-07-08; First posted 2016-10-13 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attentional Bias Modification (Experimental): ABM dot-probe task with image stimuli (faces) of three valences: positive (happy), neutral, or negative (angry and fearful). In the ABM condition, probes were located behind positive stimuli in 87 % of the trials (valid trials), as opposed to 13% with probes located behind the more negative stimuli (invalid trials). Consequently, participants should implicitly learn to deploy their attention toward positive stimuli, and in this way develop a more positive AB when completing the task.
  Interventions: Behavioral: Attentional Bias Modification
- Sham comparator (Sham Comparator): Sham condition without modification of attentional bias. These trials are identical in structure to the ABM trials with the exception that target probes replaced negative and positive images with equal frequency.
  Interventions: Behavioral: Sham Comparator

INTERVENTIONS:
Behavioral: Attentional Bias Modification — Computerized
  Arms: Attentional Bias Modification
Behavioral: Sham Comparator — Computerized
  Arms: Sham comparator

SUMMARY:
Selective biases in attention can be modified by a simple computerized technique: The Attention Bias Modification Task (ABM) pioneered by MacLeod et al. Cognitive biases may be one reason depression recurs, and altering these biases should reduce risk of recurrence. Recently, evidence has supported this hypothesis . The mechanisms by which ABM works are not well understood. More research is needed to explore how altering an implicit attentional bias can lead to changes in subjective mood. One possible explanation is that positive attentional biases are an important component of explicit methods of emotion regulation. The ability to effectively regulate one's emotions is a fundamental component of mental health and this ability is impaired in depression. It has also been shown that recovered depressed people spontaneously show a more dysfunctional pattern of emotion regulation as compared to never depressed controls. Supporting this, growing evidence implicates dysregulation of a medial/orbitofrontal circuit in mood disorders. This circuit includes the orbitofrontal cortex and anterior cingulate cortex, the ventral striatum, the ventral pallidum and medial thalamus. Components of this circuit are reciprocally connected with the amygdala, which is implicated in emotional processing in the healthy brain and dysregulated in depression. Negative emotion processing biases depend on both enhanced "bottom-up" responses to emotionally salient stimuli and reduces "top-down" cognitive control mechanisms, required to suppress responses to emotionally salient but task irrelevant information. Cognitive reappraisal and distancing are common strategies to down- or upregulate emotional responses. Reappraisal is an emotion regulation strategy that involves reinterpretation and changing the way one thinks about an event or stimulus with the goal of changing its affective impact. Distancing is a type of reappraisal that involves creating mental space between oneself and the emotional event in order to see things from a different, less self-focused perspective. It has been shown that distancing is a strategy that people can improve at over time compared to reinterpretation. The neural systems which support the explicit regulation of emotion have previously been characterized and include both lateral- and prefrontal cortex. This frontal activity is predicted to downregulate limbic circuitry involving the amygdala during passive viewing of emotional salient stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Currently no-depressed subjects with a history of major depression.

Exclusion Criteria:

* Current or past neurological illness, bipolar disorder, psychosis or drug addiction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
BOLD response in prefrontal cortical regions | Two weeks after after ABM-training
  Stronger fMRI BOLD response in prefrontal cortical regions in ABMT compared to neutral AMB placebo condition.

SECONDARY OUTCOMES:
BOLD response within the amygdala | Two weeks after ABM-training
  Lower ABM fMRI BOLD response within the amygdala in ABMT compared to neutral ABM placebo condition.
DTI | Two weeks after ABM-training
  Increased neural integrity as measured by fractional anisotropy values in the uncinate fasciculi (UF) in the active AMBT compared to neutral ABM placebo condition.
RSFC | Two weeks after ABM-training
  Increased integrity within the attentional networks at rest as measured by independent component analysis (ICA) in ABMT compared to neutral ABM training.
5-HTTLPR + A>G polymorphic variation divided by the triallelic functional "high expressive" versus "low expressive" genotype will moderate the impact from ABMT as measured by whole brain BOLD responses. | Two weeks after ABM-training
  The low expressive variant will be associated with more frontal BOLD activation and lower amygdala activation after ABMT
BDNF | Two week after ABM-training
  Brain Derived Neurotropic Factor (BDNF) val66met polymorphic variation linked to Brain Derived Neurotropic Factor (BDNF) variation will differentiate between ABMT and neutral AMB placebo as measured by fMRI whole brain BOLD responses.
Serotonergic cumulative genetic score and fMRI | Two weeks after ABM-training
  A serotonergic cumulative Genetic score, including (5-HHTLPR, HTR1A 8rs6295) and HTR 2A (rs 6311) polymorphisms will moderate the effects of ABM on fMRI BOLD signal compared to a neutral placebo condition.
Serotonergic cumulative genetic score and morphompetry | Two weeks after ABM-training
  A serotonergic cumulative Genetic score, including (5-HHTLPR, HTR1A 8rs6295) and HTR 2A (rs 6311) polymorphisms will moderate the effects of ABM on structural MRI as measured by total grey matter volume compared to a neutral placebo condition.
Serotonergic cumulative genetic score and fMRI and DTI | Two weeks after ABM-training
  A serotonergic cumulative Genetic score, including (5-HHTLPR, HTR1A 8rs6295) and HTR 2A (rs 6311) polymorphisms will moderate the effects of ABM on DTI MRI as measured by fractional anisotropy compared to a neutral placebo condition.

CONTACTS AND LOCATIONS:
Overall Officials: Nils I Landrø, phd, Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Department of Psychology, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hilland E, Landro NI ;, Harmer CJ, Browning M, Maglanoc LA, Jonassen R. Attentional bias modification is associated with fMRI response toward negative stimuli in individuals with residual depression: a randomized controlled trial. J Psychiatry Neurosci. 2020 Jan 1;45(1):23-33. doi: 10.1503/jpn.180118. PMID 31397551
- [Derived] Hilland E, Landro NI, Harmer CJ, Maglanoc LA, Jonassen R. Within-Network Connectivity in the Salience Network After Attention Bias Modification Training in Residual Depression: Report From a Preregistered Clinical Trial. Front Hum Neurosci. 2018 Dec 21;12:508. doi: 10.3389/fnhum.2018.00508. eCollection 2018. PMID 30622463